CLINICAL TRIAL: NCT01467973
Title: Gulf aCute heArt failuRe rEgistry (Gulf CARE)
Brief Title: Gulf Acute Heart Failure Registry
Acronym: GulfCARE
Status: Completed | Type: Observational
Sponsor: Gulf Heart Association (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Other Study IDs: GHA4
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Acute Heart Failure
Keywords: Heart Failure; Heart Failure, Diastolic; Heart Failure, Systolic; Middle-East
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic; Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Gulf Heart Association (GHA) sponsored Gulf acute heart failure registry (Gulf CARE)is a multinational , multicentre, prospective, observational, hospital-based registry of patients with acute heart failure(AHF) with 3 month and one year follow-up.

Study Hypothesis: Due to variations in age at presentation, risk factors for heart failure particularly high prevalence of rheumatic heart disease in certain Gulf countries, variable medical practices and heart failure management setup in the Gulf region, AHF patients in the Gulf states are expected to have different presentation and receive different management than patients in European countries resulting in different outcome. It is also hypothesized that there is considerable gap between heart failure management guidelines and clinical practices in the Gulf region.

DETAILED DESCRIPTION:
The Gulf Heart Association (GHA) initiated Gulf acute heart failure registry (Gulf CARE)is designed to assess epidemiology, clinical data, management and outcomes of AHF in six Gulf countries and whether published, professional guidelines on the diagnosis and treatment of heart failure are being applied appropriately in patients with heart failure. The registry will also provide a quantitative estimate as well as qualitative description of the hospital disease activity related to heart failure. The information gathered will identify management gaps in diagnosis and care of AHF patients that may be addressed by more effective implementation of current guidelines or development of AHF guidelines which may be appropriate to this region. Findings from this registry may help in knowing the current status of heart transplantation in the Middle-East countries as well as identify issues in establishing future heart transplant programme including selection of appropriate candidates and donors, requirements for pre- and post-transplant support.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute heart failure
* Admitted to the participating hospitals

Exclusion Criteria:

* Patients with acute heart failure who are discharged from the emergency room without admission.
* Patients transferred from non-registry hospital
* Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to various hospitals in the Middle-East with acute heart failure.
Sampling Method: Probability Sample
Enrollment: 5005 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Study of acute heart failure in the Middle-East | One year
  To describe the epidemiology, etiology, precipitating factors, demographics, clinical characteristics, management and outcome of patients admitted with acute heart failure in the Middle-East.

SECONDARY OUTCOMES:
To identify targets for the long term objectives of improving quality of care in acute heart failure patients from the Middle-East | One year
  To identify targets for the long term objectives of improving quality of care, reducing morbidity and mortality and lowering the cost of managing patients with acute heart failure in the Middle-East

CONTACTS AND LOCATIONS:
Overall Officials: Kadhim J Sulaiman, FRCPI, Principal Investigator — Royal Hospital, Muscat, Oman; Prashanth Panduranga, FRCP(Edin), Study Director — Royal Hospital
Locations (1):
- Royal Hospital, Muscat, Muḩāfaz̧at Masqaţ, Oman

REFERENCES:
- [Derived] Jan RK, Alsheikh-Ali A, Mulla AA, Sulaiman K, Panduranga P, Al-Mahmeed W, Bazargani N, Al-Suwaidi J, Al-Jarallah M, Al-Motarreb A, Salam A, Al-Zakwani I. Outcomes of guideline-based medical therapy in patients with acute heart failure and reduced left ventricular ejection fraction: Observations from the Gulf acute heart failure registry (Gulf CARE). Medicine (Baltimore). 2022 Jun 10;101(23):e29452. doi: 10.1097/MD.0000000000029452. PMID 35687781
- [Derived] Doi SA, Islam N, Sulaiman K, Alsheikh-Ali AA, Singh R, Al-Qahtani A, Asaad N, AlHabib KF, Al-Zakwani I, Al-Jarallah M, AlMahmeed W, Bulbanat B, Bazargani N, Amin H, Al-Motarreb A, AlFaleh H, Panduranga P, Shehab A, Al Suwaidi J, Salam AM. Demystifying Smoker's Paradox: A Propensity Score-Weighted Analysis in Patients Hospitalized With Acute Heart Failure. J Am Heart Assoc. 2019 Dec 3;8(23):e013056. doi: 10.1161/JAHA.119.013056. Epub 2019 Nov 29. PMID 31779564
- [Derived] Al-Zakwani I, Sulaiman K, Al-Lawati JA, Alsheikh-Ali AA, Panduranga P, Al-Habib KF, Al Suwaidi J, Al-Mahmeed W, Al-Faleh H, Elasfar A, Al-Motarreb A, Ridha M, Bulbanat B, Al-Jarallah M, Bazargani N, Asaad N, Amin H. Impact of Angiotensin Converting Enzyme Inhibitors/Angiotensin Receptors Blockers on Mortality in Acute Heart Failure Patients with Left Ventricular Systolic Dysfunction in the Middle East: Observations from the Gulf Acute Heart Failure Registry (Gulf CARE). Curr Vasc Pharmacol. 2018;16(6):596-602. doi: 10.2174/1570161115666170817164420. PMID 28820057
- [Derived] Abi Khalil C, Sulaiman K, Mahfoud Z, Singh R, Asaad N, AlHabib KF, Alsheikh-Ali A, Al-Jarallah M, Bulbanat B, AlMahmeed W, Ridha M, Bazargani N, Amin H, Al-Motarreb A, Faleh HA, Elasfar A, Panduranga P, Suwaidi JA; GULF-CARE group. Non-withdrawal of beta blockers in acute decompensated chronic and de novo heart failure with reduced ejection fraction in a prospective multicentre study of patients with acute heart failure in the Middle East. BMJ Open. 2017 Jul 9;7(7):e014915. doi: 10.1136/bmjopen-2016-014915. PMID 28694343
- [Derived] Khafaji HA, Sulaiman K, Singh R, AlHabib KF, Asaad N, Alsheikh-Ali A, Al-Jarallah M, Bulbanat B, AlMahmeed W, Ridha M, Bazargani N, Amin H, Al-Motarreb A, AlFaleh H, Elasfar A, Panduranga P, Al Suwaidi J. Clinical characteristics, precipitating factors, management and outcome of patients with prior stroke hospitalised with heart failure: an observational report from the Middle East. BMJ Open. 2015 Apr 23;5(4):e007148. doi: 10.1136/bmjopen-2014-007148. PMID 25908674